CLINICAL TRIAL: NCT06263296
Title: The Impact on Quality of Life in Individual with Burn Injury: Utilizing Smartphone Assisted Self-management Education At Aftercare
Brief Title: Smartphone Assisted Self-management Education for Adult Burn Patient At Aftercare
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Liu Siu Kwong, Associate Nurse Consultant, Department of Surgery, Principal Investigator, Queen Mary Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW 24-055
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-05

CONDITIONS: Burns; Self Efficacy; Burn Second Degree; Burns Third Degree; Quality of Life; Adherence, Treatment; Burn Injury
MeSH Terms: conditions — Burns; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: Pilot Randomized Controlled Trial
Who Masked: Participant
Masking Description: Only subject will be single blinded to the intervention provided
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional Group (Experimental): For intervention group, principal investigator will assess subject health care needs prior to intervention. Two extra sessions, 20 minutes, face to face, individual self-management education with aid of computer, track log sheet will be provided to intervention group. Concept of motivational interviewing will be incorporated as complement teaching strategy to facilitate self-management learning. Principal investigator will be responsible to deliver burn self-management education upon discharge. Intervention group will receive "Rehabilitation Booklet for Burn Patients" upon discharge. After discharge, only intervention group subject receives two sessions, 10 minutes, telephone follow up calls and five personalized chat-based messaging follow up will be provided. Besides that, self-management education information will be delivered to intervention group via instant messaging service as well.
  Interventions: Behavioral: Self Management Education
- Control Group (No Intervention): For control group, participants will receive usual care by ward nurses (provide burn discharge pamphlet upon discharge + regular plastic surgeon follow up)

INTERVENTIONS:
Behavioral: Self Management Education — Smartphone assisted self management education incorporated with the concept of motivational interviewing
  Arms: Interventional Group

SUMMARY:
Burn rehabilitation management is dependent on the patients themselves, non-treatment adherence may delay the optimal timing of burn rehabilitation and it may not be regained easily. The inevitable sequelae of increasing joint stiffness and tethered soft-tissue glide become more devastating over time. It has a major impact on clinical outcomes such as scarring, deformity and dysfunction, which result in lower quality of life compared to general population

There is a growing body of research on patient-centered interventions including the concept of self-management. Such phenomenon is consistent with burn patients' needs at aftercare. The proposed smartphone self-management program is to change the paradigm from paternalistic to collaborative relationship. Self-management is to build up patient equipping ability in problem solving, decision making, and appropriate use of resources and has led to improved patient engagement, adherence, and better quality of care.

The investigators hypothesize that, upon intervention completion and compared with the control group, burn patients in the intervention group will report:

1. Higher level of health-related quality of life,
2. Higher level of self-efficacy
3. Higher level of score in Burn Rehabilitation Knowledge
4. Lower pain level, as measured by Numeric Pain Rating Scale; and
5. Lower level of itchiness

The desired smart phone assisted self-management intervention will be carried out by principal investigator to selected adult burn patients before discharge and post discharge period. Before discharge, ward nurses will provide discharge pamphlet and individual face to face education to both groups as usual care. After discharge, instant messaging supportive enquiry service will be provided to both groups via smartphone apps.

For intervention group, principal investigator will assess subject health care needs prior to intervention. Two extra sessions, 20 minutes, face to face, individual self-management education with aid of computer, track log sheet will be provided to intervention group. Concept of motivational interviewing will be incorporated as complement teaching strategy to facilitate self-management learning. Principal investigator will be responsible to deliver burn self-management education upon discharge. Intervention group will receive "Rehabilitation Booklet for Burn Patients" upon discharge. After discharge, only intervention group subject receives two sessions, 10 minutes, telephone follow up calls and five personalized chat-based messaging follow up will be provided. Besides that, self-management education information will be delivered to intervention group via instant messaging service as well. Ad-hoc instant messaging support will be provided to both groups if required.

DETAILED DESCRIPTION:
Due to the advancement of medical treatment, burn-related mortality has been reduced especially in developed countries . Long-term undesirable impacts such as wound problems, skin care, exercise training, scar management, psychological and social problems have been detected in both major and non-major burns (less than 20% total body surface area (TBSA). The focus of burn care is shifted not only acute care but also rehabilitation.

Burn rehabilitation management is dependent on the patients themselves, non-treatment adherence may delay the optimal timing of burn rehabilitation and it may not be regained easily. The inevitable sequelae of increasing joint stiffness and tethered soft-tissue glide become more devastating over time. It has a major impact on clinical outcomes such as scarring, deformity and dysfunction, which result in lower quality of life compared to general population

There is a growing body of research on patient-centered interventions including the concept of self-management. Such phenomenon is consistent with burn patients' needs at aftercare. The proposed smartphone self-management program is to change the paradigm from paternalistic to collaborative relationship. Self-management is to build up patient equipping ability in problem solving, decision making, and appropriate use of resources and has led to improved patient engagement, adherence, and better quality of care.

The investigators hypothesize that, upon intervention completion and compared with the control group, burn patients in the intervention group will report:

1. Higher level of health-related quality of life,
2. Higher level of self-efficacy
3. Higher level of score in Burn Rehabilitation Knowledge
4. Lower pain level, as measured by Numeric Pain Rating Scale; and
5. Lower level of itchiness

The desired smart phone assisted self-management intervention will be carried out by principal investigator to selected adult burn patients before discharge and post discharge period.

Before discharge, ward nurses will provide discharge pamphlet and individual face to face education to both groups as usual care.

After discharge, instant messaging supportive enquiry service will be provided to both groups via smartphone apps.

For intervention group, principal investigator will assess subject health care needs prior to intervention. Two extra sessions, 20 minutes, face to face, individual self-management education with aid of computer, track log sheet will be provided to intervention group. Concept of motivational interviewing will be incorporated as complement teaching strategy to facilitate self-management learning.

Principal investigator will be responsible to deliver burn self-management education upon discharge. Intervention group will receive "Rehabilitation Booklet for Burn Patients" upon discharge.

After discharge, only intervention group subject receives two sessions, 10 minutes, telephone follow up calls and five personalized chat-based messaging follow up will be provided. Besides that, self-management education information will be delivered to intervention group via instant messaging service as well. Ad-hoc instant messaging support will be provided to both groups if required.

ELIGIBILITY:
Inclusion Criteria:

* Chinese adult aged above 18 years old
* Hospitalized burn patient
* Adult who can understand Cantonese
* Superficial partial thickness burn: TBSA >10%
* Deep partial thickness burn or full thickness burn: TBSA > 5%

Exclusion Criteria:

* Inhalation injury solely
* Sustained burn injury due to self-injury
* Diagnosed psychiatric illness with or without medication
* Client who is unable to communicate via instant messaging apps

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-10 (Actual); Primary Completion 2025-08-28 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Disease Specific Quality of life at Week 4 & Week 12 | Baseline and Week 4; Week 12
  Burn Specific Health Scale-Brief (BSHS-B) Taiwanese version (40-items, Appendix 7) will be used to quantify the recovery of quality of life (QoL) among burn survivor in general, physical, mental, and social health aspects. Responses are measured on a 5-point scale ranging from 0 ("extreme") to 4 ("none at all"). The total (BSHS-B score is the sum of the subscale scores (range: 0-160), with a higher score indicating better quality of life post burn injury.
Change from Baseline in the Generic Quality of life at Week 4 & Week 12 | Baseline and Week 4; Week 12
  5Q-5D-5L Hong Kong- Traditional Chinese version (Appendix 8) ls used to measure the generic health-related quality of life (HRQoL) among subjects. It has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) with five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). The digits for the five dimensions can be combined in a 5-digit code that describes the respondent's health state.
Change from Baseline in the Burn Rehabilitation Knowledge Questionnaire | Baseline and Week 4
  The Burn Rehabilitation Knowledge Questionnaire is developed by the principal investigator after reviewing the relevant and recent international scientific literature to identify patients' learning needs and essential concept in facilitating burn rehabilitation. This questionnaire consisted of twenty-four multiple choice questions covering three well-defined areas: general knowledge about burns (8 items), rehabilitation modalities (8 items), and burns related healthy lifestyle modifications (8 items). The total scores were computed out of (24 grades). A higher score indicated better knowledge in burn rehabilitation.

SECONDARY OUTCOMES:
Change from Baseline in the Self efficacy at Week 4 & Week 12 | Baseline and Week 4; Week 12
  Chinese Adaptation of the General Self-Efficacy Scale (C-GSE, 10 items, Appendix 9) will be used to measure the sense of self efficacy of the patients. The General Self-Efficacy Scale is correlated to emotion, optimism, work satisfaction. Negative coefficients were found for depression, stress, health complaints, burnout, and anxiety. Responses are measured on a 4-point scale ranging from 1 ("Not at all") to 4 ("Exactly True"). The total GSE score is the sum of the subscale scores (range: 10-40), with a higher score indicating more self-efficacy.
Change from Baseline in the Itchiness of life at Week 4 & Week 12 | Baseline and Week 4; Week 12
  5D itch score(5D-IS)- Chinese version (Appendix 10) will be used to measure severity of itchiness in five dimensions which are degree, duration, direction, disability and distribution. the first four domains were measured on a five-point Likert scale. The distribution domain included 16 potential locations of itch, the more itchy area, the higher score will be obtained in this domain. Responses are measured on a 5-point scale ranging from 1 to 5 ranged between 5 (no pruritus) and 25 (most severe pruritus).
Change from Baseline in the Pain level at Week 4 & Week 12 | Baseline and Week 4; Week 12
  Numeric Pain Rating Scale (NPRS) will be used to measure the subjective intensity of pain. Responses are measured on a 11-point scale ranging from 0 ("no pain") to 10 ("the most intense pain imaginable").

OTHER OUTCOMES:
Percentage in the Burn related out-patient clinic attendance | Week 4; Week 12
  Burn related out-patient clinic attendance including doctor, nurse, allied health after discharge will be traced back within three months.

CONTACTS AND LOCATIONS:
Locations (1):
- LIU Siu Kwong, Hong Kong, China

REFERENCES:
- [Background] Procter F. Rehabilitation of the burn patient. Indian J Plast Surg. 2010 Sep;43(Suppl):S101-13. doi: 10.4103/0970-0358.70730. PMID 21321643
- [Background] Spronk I, Legemate C, Oen I, van Loey N, Polinder S, van Baar M. Health related quality of life in adults after burn injuries: A systematic review. PLoS One. 2018 May 24;13(5):e0197507. doi: 10.1371/journal.pone.0197507. eCollection 2018. PMID 29795616
- [Background] Esselman PC. Burn rehabilitation: an overview. Arch Phys Med Rehabil. 2007 Dec;88(12 Suppl 2):S3-6. doi: 10.1016/j.apmr.2007.09.020. PMID 18036978
- [Background] Smolle C, Cambiaso-Daniel J, Forbes AA, Wurzer P, Hundeshagen G, Branski LK, Huss F, Kamolz LP. Recent trends in burn epidemiology worldwide: A systematic review. Burns. 2017 Mar;43(2):249-257. doi: 10.1016/j.burns.2016.08.013. Epub 2016 Sep 3. PMID 27600982
- [Background] Barrett LW, Fear VS, Waithman JC, Wood FM, Fear MW. Understanding acute burn injury as a chronic disease. Burns Trauma. 2019 Sep 16;7:23. doi: 10.1186/s41038-019-0163-2. eCollection 2019. PMID 31534977